CLINICAL TRIAL: NCT00723775
Title: Phase I, Open Label Drug-drug Interaction Study in Healthy Volunteers to Evaluate the Effect of KALETRA (Lopinavir-ritonavir) on GSK706769 Pharmacokinetics and to Evaluate the Pharmacokinetics of a New Oral Formulation of GSK706769
Brief Title: GSK706769/KALETRA Drug-drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRR110744
Record Dates: First submitted 2008-07-28; First posted 2008-07-29 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: KALETRA; GSK706769; HIV; healthy volunteers
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — lopinavir-ritonavir drug combination

ARMS (2):
- Part 1 (Other): GSK706769 new vs. current formulation; GSK706769 alone vs. GSK706769 plus Kaletra
  Interventions: Drug: GSK706769 & KALETRA
- Part 2 (Other): GSK706769 alone for 10 days; GSK706769 + Kaletra for 14 days
  Interventions: Drug: GSK706769 & KALETRA

INTERVENTIONS:
Drug: GSK706769 & KALETRA — GSK706769 alone and GSK706769 + Kaletra

SUMMARY:
To compare plasma GSK706769 PK following repeat administration of GSK706769 QD with and without KALETRA (LPV 400 mg/RTV 100mg) q12h

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male or female between 18 and 50 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:
* Is pre-menopausal females with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries), or hysterectomy;
* Is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 mlU/ml is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt, HRT should be discontinued for 2 weeks and then the subject rescreened, as HRT can suppress FSH. Following confirmation of their post-menopausal status, they can resume use of HRT.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of medication.
* Body weight >= 50 kg (110 lbs.) for men and >=45 kg (99 lbs) for women and BMI within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >14 drinks/week for men or >7 drinks/week for women.

Note: One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatic diseases.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* The subject has received GSK706769 in a previous clinical trial.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.

Note: "Study" or "investigational" drugs include GSK706769 or Kaletra

- Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Note: this does not include plasma donation.

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG per protocol.
* Exclusion Criteria for 24-Hour Screening Holter per protocol (conducted only if telemetry is warranted from findings on telemetry from an ongoing repeat dose study):

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-07-24 (Actual); Primary Completion 2008-11-08 (Actual); Study Completion 2008-11-08 (Actual)

PRIMARY OUTCOMES:
GSK706769 PK | Part 1: 4 days; Part 2; 25 days

SECONDARY OUTCOMES:
GSK706769 safety parameters, including adverse events, clinical laboratory, ECG, and vital signs assessments. | Part 1: 4 days; Part 2; 25 days
Plasma GSK706769 AUC(0-∞), AUC(0-t), and Cmax following a single dose of GSK706769 50mg and following combined administration of a single dose of GSK706769 50mg with a single dose of LPV 400mg/RTV 100mg. | Part 1: 4 days; Part 2; 25 days
Plasma metabolite GSK1996847 AUC(0-∞), AUC(0-t), and Cmax following a single dose of GSK706769 50mg and following combined administration of a single dose of GSK706769 50mg with a single dose of LPV 400mg/RTV 100mg. | Part 1: 4 days; Part 2; 25 days
Metabolite GSK1996847 AUC(0-t) and Cmax following repeat dose administration of GSK706769 QD for 10 days and following coadministration with Kaletra (LPV 400mg/RTV 100mg) q12h for 14 days. | Part 1: 4 days; Part 2; 25 days
Plasma protein and mRNA expression levels of biomarkers before and after administration of GSK706769 QD for 5 days. | Part 1: 4 days; Part 2; 25 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study CRR110744 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/CRR110744?search=study&search_terms=CRR110744#rs